CLINICAL TRIAL: NCT01502982
Title: CHOEP-14 + Rituximab With CNS Prophylaxis in Patients Less Than 65 Years With Diffuse Large B-Cell Lymphoma/Follicular Lymphoma Grade III, Stage II-IV With Risk Factors (Age Adjusted IPI) ≥ 2. A Phase II Study
Brief Title: Dose Dense Chemotherapy and Rituximab for Young High Risk Diffuse Large B-Cell Lymphoma Patients (CRY-04)
Acronym: CRY-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Lymphoma Group (Network)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG-LBC-04; 2004-003075-37 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2012-01-02 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; high risk; young
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemoimmunotherapy (Experimental)
  Interventions: Drug: R-CHOEP14x6+HD-AraC+HD-Mtx

INTERVENTIONS:
Drug: R-CHOEP14x6+HD-AraC+HD-Mtx — rituximab 375 mg/m2 day 1 cyclophosphamide 750 mg/m2 day 1 doxorubicin 50 mg/m2 day 1 vincristine 1.4 mg/m2 day 1 etoposide 100mg/m2 days 1,2,3 Prednison 100 mg days 1,2,3,4,5 cycle repeated six times every two weeks followed by HD-AraC 3g/m2x4 and HD-mtx 3 g/m2 HD-AraC 3g/m2x4 times every 12 h
  Other Names: R-CHOEP14x6; HD-MTXx1; HD-AraCx1

SUMMARY:
The purpose is to test whether dose densified chemoimmunotherapy followed by central nervous system (CNS) prophylaxis for young high risk diffuse large B-cell lymphoma (DLBCL) patients is feasible and could improve time to treatment failure and reduce the risk of CNS relapses. Six courses of rituximab-cyclophosphamide-doxorubicin-etoposide-vincristine-prednison (R-CHOEP) given in two weeks intervals with the support of G-CSF is followed by one course of high dose methotrexate (HD-MTX) and high dose cytarabine (HD-Ara-C). The results will be compared to a historical Nordic study.

DETAILED DESCRIPTION:
Pathology:

Patients may be included on the bases of the histological diagnosis of the local pathologist. The specimen will be reviewed by a central pathologist in each country

Treatment:

All patients receive CHOEP-14 with rituximab x 6 with the support of G-CSF followed by high dose cytarabine i.v. and high dose methotrexate i.v.Intrathecal (i.t.) CNS prophylaxis in combination with chemotherapy is not to be given, but i.t. methotrexate may be given once after initial liquid sampling. Radiotherapy will be given at the discretion of the individual centres.

Investigations before, during and after treatment:

The disease status will be assessed prior to treatment start, after 3 cycles of CHOEP + rituximab and after completion of the treatment schedule. Positron Emission Tomography (PET) using F18 deoxyglucose may be performed after fulfillment of treatment. Persistent, suspected lymphoma tissue should whenever possible be confirmed with a biopsy, otherwise the patient will be regarded as PR and second line therapy will be considered (see schematic outline).

Clinical and radiological (CT) assessment are performed at pretreatment and subsequently on sites initially involved, and bone marrow biopsy if initially involved

* After the 3rd course
* After the last course (within one month) of chemotherapy (biopsy if indicated)
* After radiotherapy (for patient given radiotherapy as part of the primary treatment)

Clinical follow-up:

* 4x per year during the first and second year of follow-up
* 2x per year during the third, fourth and fifth year of follow-up

Radiological investigations at follow up:

-CT after 6, 12 and 24 months of sites initially involved. CT abdomen in all cases after 12 and 24 months. X-ray of the thorax (if CT thorax is performed) after 6, 12 and 24 months

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 - < 65 years.
2. Histology verified according to the WHO classification and with CD20 positivity by immunhistochemistry or flow cytometry:

   * Diffuse large B-cell lymphomas with subgroups except posttransplantation-, Burkitt-like- and primary CNS lymphomas and cases with leptomeningeal lymphoma involvement. Morphologically discordant lymphomas (most often follicular lymphoma and diffuse large cell B-cell lymphoma in different biopsy specimens, e.g. lymphatic gland and bone marrow) and transformed lymphomas are not to be included.
   * Follicular lymphomas grade III The diagnosis made by the local pathologist of the participating centre will be accepted for registration
3. Patients in at least stage II with age adjusted IPI score of 2 or 3:

   Stage III /IV and elevated LDH and/or WHO performance status 2 - 3 Stage II and elevated LDH and WHO performance status 2 - 3.
4. Previously untreated.
5. Performance status < 4 (Appendix 2).
6. Written informed consent

Exclusion Criteria:

1. Severe cardiac disease: cardiac function grade 3-4 (Appendix 2) or Left Ventricular Ejection Fraction (LVEF) < 45% (based on MUGA scintigraphy or echo Doppler cardiography).
2. Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule.
3. Pregnancy.
4. Men and women of reproductive potential not agreeing to use an acceptable method of birth control during treatment and for six months after completion of treatment.
5. Patients with other severe medical problems and with an expected short survival for non-lymphoma reasons.
6. Known HIV positivity.
7. Present or previous cancer except basal cell carcinoma and cervical carcinoma in situ.
8. Uncontrolled infectious disease.
9. Psychiatric or mental disorder which make the patient unable to give an informed consent and/or adhere to the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2004-11; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | 5 years
  Interval between the registration date and the date of documented progression or lack of response, first relapse, death for any reason or discontinuation/change of therapy because of toxicity, whichever occurs first. Otherwise, patients will be censored at the last date they were known to be alive. For patients not responding at any time point on study treatment, TTF is defined as 1 day.

SECONDARY OUTCOMES:
Number of participants with adverse events | Treatment period (5 years)
  Grade 2-4 hematological and non-hematological adverse events according to the WHO Common Toxicity Criteria as specified in the protocol
Clinical response rate | Treatment period (5 years)
  Number of patients with complete and partial responses, stable or progressive disease after 3 courses and the end of treatment period
Time to progression | 5 years
  Time from registration to the date of disease progression. Otherwise, the patients are censored at the last date of follow up. Patients still alive in a complete response or lost to follow-up are censored at the last date they were known to be alive. Patients who die due to causes other than lymphoma are censored at the date of death
Overall survival | 5 years
  Time from the registration date to the date of death. Patients still alive or lost to follow-up are censored at the last date they were known to be alive.
Incidence of CNS relapse | Treatment period (5 years)
Molecular factors important for clinical outcome | Treatment period (5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Holte, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (4):
- Odense University Hospital, Odense, Denmark
- Helsinki University central Hospital, Helsinki, Finland
- Oslo University Hospital, Oslo, Norway
- Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Autio M, Leivonen SK, Bruck O, Mustjoki S, Meszaros Jorgensen J, Karjalainen-Lindsberg ML, Beiske K, Holte H, Pellinen T, Leppa S. Immune cell constitution in the tumor microenvironment predicts the outcome in diffuse large B-cell lymphoma. Haematologica. 2021 Mar 1;106(3):718-729. doi: 10.3324/haematol.2019.243626. PMID 32079690
- [Derived] Taskinen M, Louhimo R, Koivula S, Chen P, Rantanen V, Holte H, Delabie J, Karjalainen-Lindsberg ML, Bjorkholm M, Fluge O, Pedersen LM, Fjorden K, Jerkeman M, Eriksson M, Hautaniemi S, Leppa S. Deregulation of COMMD1 is associated with poor prognosis in diffuse large B-cell lymphoma. PLoS One. 2014 Mar 13;9(3):e91031. doi: 10.1371/journal.pone.0091031. eCollection 2014. PMID 24625556
- [Derived] Holte H, Leppa S, Bjorkholm M, Fluge O, Jyrkkio S, Delabie J, Sundstrom C, Karjalainen-Lindsberg ML, Erlanson M, Kolstad A, Fossa A, Ostenstad B, Lofvenberg E, Nordstrom M, Janes R, Pedersen LM, Anderson H, Jerkeman M, Eriksson M. Dose-densified chemoimmunotherapy followed by systemic central nervous system prophylaxis for younger high-risk diffuse large B-cell/follicular grade 3 lymphoma patients: results of a phase II Nordic Lymphoma Group study. Ann Oncol. 2013 May;24(5):1385-92. doi: 10.1093/annonc/mds621. Epub 2012 Dec 17. PMID 23247661
- [Derived] Riihijarvi S, Nurmi H, Holte H, Bjorkholm M, Fluge O, Pedersen LM, Rydstrom K, Jerkeman M, Eriksson M, Leppa S. High serum vascular endothelial growth factor level is an adverse prognostic factor for high-risk diffuse large B-cell lymphoma patients treated with dose-dense chemoimmunotherapy. Eur J Haematol. 2012 Nov;89(5):395-402. doi: 10.1111/ejh.12005. Epub 2012 Sep 14. PMID 22882209
- See also: Nordic Lymphoma Group — http://www.nordic-lymphoma.org/